CLINICAL TRIAL: NCT04223635
Title: An Open-label, Single-dose Study to Assess the Pharmacokinetics of Pexidartinib in Subjects With Moderate Hepatic Impairment Compared to Healthy Subjects
Brief Title: Study of Pexidartinib in Participants With Moderate Hepatic Impairment Compared With Healthy Participants
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PL3397-A-U129
Record Dates: First submitted 2020-01-06; First posted 2020-01-10 (Actual); Results first posted 2021-06-07 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Moderate Hepatic Impairment
Keywords: Moderate hepatic impaired; Healthy subjects; Pexidartinib; Clinical pharmacology study; Tenosynovial giant cell tumor (TGCT)
MeSH Terms: conditions — Giant Cell Tumor of Tendon Sheath | interventions — pexidartinib

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Hepatic impaired (Experimental): Participants with moderate hepatic impairment who will receive a single oral dose of pexidartinib.
  Interventions: Drug: Pexidartinib
- Healthy controls (Experimental): Sex-, age-, and weight-matched healthy participants who will receive a single oral dose of pexidartinib.
  Interventions: Drug: Pexidartinib

INTERVENTIONS:
Drug: Pexidartinib — Single, 200-mg capsule will be administered orally on Day 1 with 240 mL of water, following an overnight fast of at least 10 hours.

SUMMARY:
The pharmacokinetics of a single dose of pexidartinib was investigated in participants with impaired hepatic function and compared with healthy control participants with normal hepatic function.

DETAILED DESCRIPTION:
Pexidartinib is an orally administered tyrosine kinase inhibitor, currently approved in the US for the treatment of adult patients with symptomatic tenosynovial giant cell tumor (TGCT) associated with severe morbidity or functional limitations and not amenable to improvement with surgery.

The primary objective of this study is to determine the plasma pharmacokinetics (PK) of pexidartinib after a single oral dose of 200 mg in participants with moderate hepatic impairment (HI) as defined by National Cancer Institute Organ Dysfunction Working Group (NCI-ODWG) criteria compared to the healthy controls participants with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

• Screening: Male and female participants, 18 y to 75 years of age, inclusive, with body mass index (BMI) 18 kg/m^2 to 40 kg/m^2, inclusive at Screening.

Participants with hepatic impairment (HI) are required to have:

* Documented history of chronic liver disease diagnosed by ultrasonography, computed tomography scan, liver biopsy, or magnetic resonance imaging or history of chronic (>6 months) hepatitis B virus or hepatitis C virus infection.
* Moderate HI as assessed by the National Cancer Institute-Organ Dysfunction Working Group (NCI-ODWG) criteria (total bilirubin [TBIL] >1.5 to 3x upper limit of normal [ULN]) not due to Gilbert's syndrome.
* Normal or nonclinically relevant findings at physical examination and normal limits or nonclinically relevant deviations in clinical laboratory evaluations, with exception of findings that in the opinion of investigator are consistent with participant's HI.
* Clinical stability in the opinion of the investigator.
* Female participants (both, healthy and HI participants) who are of non-childbearing potential must be:

  * Surgically sterile (ie, bilateral tubal ligation or removal of both ovaries and/or uterus at least 6 months prior to dosing, or Essure® with hysterosalpingogram [documentation to confirm tubal occlusion 12 weeks after procedure]).
  * Naturally postmenopausal (spontaneous cessation of menses) for at least 12 consecutive months prior to dosing, confirmed by follicle stimulating hormone (FSH) or estradiol testing.
* Female participants (both, healthy and HI subjects) who are of childbearing potential must agree to barrier method of contraceptive therapy or refrain from sexual intercourse to prevent pregnancy until 1 month post dose. If the participant is on oral contraceptive, the participant needs to use the barrier method in addition to oral contraceptive. Female participants must refrain from breastfeeding for at least 2 weeks post dose.
* Male participants (both, healthy and HI subjects) must surgically sterile or agree to use double barrier methods of contraception from Check-in until 1 month after the dose of pexidartinib. Also, male participants must not donate sperm from Check-in until 1 month after pexidartinib administration.

Exclusion Criteria:

* Clinically relevant abnormal history, physical findings, ECG, or laboratory values at the Screening assessment that could interfere with the objectives of the study or the safety of the participant
* Participants with primary biliary cirrhosis or primary sclerosing cholangitis
* Concomitant medication (moderate or strong inhibitor or inducer of CYP3A4 [eg, itraconazole, rifampin], CYP2C9 [eg, fluconazole, carbamazepine] and uridine 5'-diphospho-glucuronosyltransferase (UGT) [eg, probenecid, rifampin]) within 2 weeks before dosing and throughout study
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (with the exception of appendectomy, hernia repair, and/or cholecystectomy)
* Presence or history of severe adverse reaction to any drug (except penicillin)
* A positive drugs of abuse screen (unless the drug is medically prescribed by a licensed health care provider) or alcohol breath test at Screening or at Check-in on Day -2 or a participant who will not agree to smoke ≤10 cigarettes or equivalent per day from Screening up to Enrollment, and is unable to be restricted to ≤5 cigarettes per day and for 6 hours post dose during their period of residence in the clinical unit
* Concomitant use of medications known to affect the elimination of serum creatinine (eg, trimethoprim or cimetidine) and inhibitors of renal tubular secretion (eg, probenecid) within 60 days of Day -2
* History or presence of an abnormal ECG, which, in the investigator's opinion, is clinically significant and/or a QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥450 milliseconds (ms) and ≥470 ms for healthy male and female participants, respectively, and >500 ms for participants with HI at Screening
* Consumption of alcohol-within 72 hours prior to Check-in and caffeine-containing beverages within 48 hours prior to Check-in and during confinement
* Consumption of more than 28 units of alcohol per week for males or 14 units of alcohol per week for females, where 1 unit of alcohol equals one-half pint of beer, 4 ounces (oz) of wine, or 1 oz of spirits, or significant history of alcoholism or drug/chemical abuse within the last 2 years
* Positive serology for HBsAg and anti-hepatitis C virus (HCV) (healthy participants), hepatitis A virus (HAV) immunoglobulin M, or anti-HIV Type 1 and Type 2 (all participants)
* Loss of more than 450 mL blood during the 3 months before the trial (eg, as a blood donor)
* Current enrollment in or have not yet completed at least 30 days or 5 elimination half-lives, whichever is longer, since receiving an investigational device or product, or receipt of other investigational agents within 30 days of pexidartinib

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2020-10-02 (Actual); Study Completion 2020-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Leader, Study Director — Daiichi Sankyo
Locations (2):
- United States (2):
  - Clinical Pharmacology of Miami, LLC., Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Zahir H, Greenberg J, Hsu C, Marbury TC, Lasseter KC, Xu LA, Tap WD, Healey JH, Stacchiotti S, LaCreta F. Effect of Mild and Moderate Hepatic Impairment (Defined by Child-Pugh Classification and National Cancer Institute Organ Dysfunction Working Group Criteria) on Pexidartinib Pharmacokinetics. J Clin Pharmacol. 2022 Aug;62(8):992-1005. doi: 10.1002/jcph.2042. Epub 2022 Mar 31. PMID 35247274

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 16 participants who met all inclusion criteria and no exclusion criteria were enrolled from 07 Jan 2020 to 02 Oct 2020 at 2 clinics in the United States.
Groups:
- Normal HF: Healthy matched participants with normal hepatic function (HF) who received 200mg pexidartinib on Day 1 with 240 mL water. Participants fasted for at least 10 hours(h) before pexidartinib dosing and continued to fast for at least 4h after pexidartinib administration.
- Moderate HI: Participants with moderate HI who received 200mg pexidartinib on Day 1 with 240 mL water. Participants fasted for at least 10 hours(h) before pexidartinib dosing and continued to fast for at least 4h after pexidartinib administration. Moderate hepatic impairment (HI) was assessed by National Cancer Institute - Organ Dysfunction Working Group (NCI-ODWG).
Period: Overall Study
Arm/Group | Normal HF | Moderate HI
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were assessed using the Safety Analysis Set.
Groups:
- Normal HF: Healthy matched participants with normal HF who received 200mg pexidartinib on Day 1 with 240 mL water. Participants fasted for at least 10h before pexidartinib dosing and continued to fast for at least 4h after pexidartinib administration.
- Moderate HI: Participants with moderate HI who received 200mg pexidartinib on Day 1 with 240 mL water. Participants fasted for at least 10h before pexidartinib dosing and continued to fast for at least 4h after pexidartinib administration. Moderate hepatic impairment (HI) was assessed by National Cancer Institute - Organ Dysfunction Working Group (NCI-ODWG).
- Total: Total of all reporting groups
Arm/Group | Normal HF | Moderate HI | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 7 | 13
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (6.69) | 59.4 (4.34) | 58.8 (5.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 6 | 7 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kilogram] | 86.30 (13.49) | 78.13 (14.83) | 82.21 (14.33)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of Pexidartinib Following a Single Dose in Participants With Moderate Hepatic Impairment Compared to Healthy Participants
Description: Maximum Plasma Concentration (Cmax) is defined as the maximum observed plasma concentration and was calculated using non-compartmental analysis.
Time Frame: Pre-dose (within 60 minutes prior to dosing) and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144, and 168 hours post-dose
Population: Pharmacokinetic parameter was assessed using the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Normal HF | Moderate HI
Number analyzed (Participants) | 8 | 8
ng/mL | 1420 (738) | 1250 (556)
Statistical Analysis 1: Comparison: Normal HF vs Moderate HI; Test type: Other — Least squares (LS) means were calculated from an analysis of variance (ANOVA) model on log-transformed scale. The LS means for each treatment were back transformed from the log scale to provide estimates of the geometric means (GMS). The ratio (%) of GMS was calculated and 90% Confidence Interval (CIs) for the ratio (%) of GMS were presented; Ratio (%) of Geometric LS Mean = 92.60, 90% CI 2-sided [54.38 to 157.69] — For the comparison, moderate HI represents the numerator and normal HF represents the denominator

2. Primary Outcome: Time of Maximum Plasma Concentration (Tmax) of Pexidartinib Following a Single Dose in Participants With Moderate Hepatic Impairment Compared to Healthy Participants
Description: Time of Maximum Plasma Concentration (Tmax) is defined as the time of maximum observed plasma concentration and was calculated using non-compartmental analysis.
Time Frame: as for outcome 1
Population: Pharmacokinetic parameter was assessed using the Pharmacokinetic Analysis Set.
Measure: Median (Full Range); unit: hours
Arm/Group | Normal HF | Moderate HI
Number analyzed (Participants) | 8 | 8
hours | 1.9 [1.5 to 4.5] | 2.5 [2.0 to 3.0]

3. Primary Outcome: Area Under the Plasma Concentration-Time Curve up to the Last Quantifiable Concentration Post-Dose (AUClast) of Pexidartinib Following a Single Dose in Participants With Moderate Hepatic Impairment Compared to Healthy Participants
Description: Area Under the Plasma Concentration-Time Curve up to the Last Quantifiable Concentration Post-Dose (AUClast) is defined as AUC from time 0 to the last measurable concentration, as calculated by the linear up-log down trapezoidal method and was calculated using non-compartmental analysis.
Time Frame: as for outcome 1
Population: Pharmacokinetic parameter was assessed using the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng•h/mL
Arm/Group | Normal HF | Moderate HI
Number analyzed (Participants) | 8 | 8
ng•h/mL | 26500 (12200) | 38600 (16200)
Statistical Analysis 1: Comparison: Normal HF vs Moderate HI; Test type: Other — Least squares means were calculated from an analysis of variance (ANOVA) model on log-transformed scale. The LS means for each treatment were back transformed from the log scale to provide estimates of the geometric means (GMS). The ratio (%) of GMS was calculated and 90% CIs for the ratio (%) of GMS were presented; Ratio (%) of Geometric Least Square Mean = 147.17, 90% CI 2-sided [95.39 to 227.07] — For the comparison, moderate HI represents the numerator and normal HF represents the denominator

4. Primary Outcome: Area Under the Plasma Concentration-Time Curve up to Infinity (AUCinf ) of Pexidartinib Following a Single Dose in Participants With Moderate Hepatic Impairment Compared to Healthy Participants
Description: Area Under the Plasma Concentration-Time Curve up to Infinity (AUCinf ) is defined as area under the plasma concentration-time curve from the time of dosing extrapolated to infinity and was calculated using non-compartmental analysis.
Time Frame: as for outcome 1
Population: The pharmacokinetic parameter of Area Under the Plasma Concentration-Time Curve up to Infinity was assessed using the Pharmacokinetic Analysis Set except for 1 participant that did not meet the protocol inclusion criteria for this analysis.
Measure: Mean (Standard Deviation); unit: ng•h/mL
Arm/Group | Normal HF | Moderate HI
Number analyzed (Participants) | 8 | 7
ng•h/mL | 27300 (12400) | 38900 (17600)
Statistical Analysis 1: Comparison: Normal HF vs Moderate HI; Test type: Other — [test comment as in outcome 3, analysis 1]; Ratio (%) of Geometric Least Square Mean = 142.87, 90% CI 2-sided [91.21 to 223.79] — For the comparison, moderate HI represents the numerator and normal HF represents the denominator

5. Primary Outcome: Elimination Rate Constant (Kel) of Pexidartinib Following a Single Dose in Participants With Moderate Hepatic Impairment Compared to Healthy Participants
Description: Elimination Rate Constant (Kel) is defined as elimination rate constant and was calculated using non-compartmental analysis.
Time Frame: as for outcome 1
Population: The pharmacokinetic parameter of Elimination Rate Constant was assessed using the Pharmacokinetic Analysis Set except for 1 participant that did not meet the protocol inclusion criteria for this analysis..
Measure: Mean (Standard Deviation); unit: fraction per hour
Arm/Group | Normal HF | Moderate HI
Number analyzed (Participants) | 8 | 7
fraction per hour | 0.02294 (0.002072) | 0.019784 (0.0042775)

6. Primary Outcome: Terminal Elimination Half-Life (t1/2) of Pexidartinib Following a Single Dose in Participants With Moderate Hepatic Impairment Compared to Healthy Participants
Description: Terminal Elimination Half-Life (t1/2) is defined as terminal elimination half-life and was calculated using non-compartmental analysis.
Time Frame: as for outcome 1
Population: The pharmacokinetic parameter of Terminal Elimination Half-Life was assessed using the Pharmacokinetic Analysis Set except for 1 participant that did not meet the protocol inclusion criteria for this analysis.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Normal HF | Moderate HI
Number analyzed (Participants) | 8 | 7
hours | 30.4 (2.58) | 36.5 (8.05)

7. Primary Outcome: Total Apparent Clearance (CL/F) of Pexidartinib Following a Single Dose in Participants With Moderate Hepatic Impairment Compared to Healthy Participants
Description: Total Apparent Clearance (CL/F) is defined as total apparent clearance and was calculated using non-compartmental analysis.
Time Frame: as for outcome 1
Population: The pharmacokinetic parameter of Total Apparent Clearance was assessed using the Pharmacokinetic Analysis Set except for 1 participant that did not meet the protocol inclusion criteria for this analysis.
Measure: Mean (Standard Deviation); unit: liters per hour
Arm/Group | Normal HF | Moderate HI
Number analyzed (Participants) | 8 | 7
liters per hour | 9.046 (5.1294) | 6.270 (3.2935)

8. Primary Outcome: Volume of Distribution in the Terminal Phase (Vz/F) Following a Single Dose in Participants With Moderate Hepatic Impairment Compared to Healthy Participants
Description: Volume of Distribution in the Terminal Phase (Vz/F) is defined as volume of distribution in the terminal phase and was calculated using non-compartmental analysis.
Time Frame: as for outcome 1
Population: The pharmacokinetic parameter of Volume of Distribution in the Terminal Phase was assessed using the Pharmacokinetic Analysis Set except for 1 participant that did not meet the protocol inclusion criteria for this analysis.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Normal HF | Moderate HI
Number analyzed (Participants) | 8 | 7
liters | 391.6 (205.29) | 343.0 (238.12)

9. Secondary Outcome: Maximum Plasma Concentration (Cmax) of ZAAD-1006a Metabolite Following a Single Dose of Pexidartinib in Participants With Moderate Hepatic Impairment Compared to Healthy Participants
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Pharmacokinetic parameter was assessed using the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Normal HF | Moderate HI
Number analyzed (Participants) | 8 | 8
ng/mL | 1720 (950) | 1250 (766)

10. Secondary Outcome: Maximum Plasma Concentration (Tmax) of ZAAD-1006a Metabolite Following a Single Dose of Pexidartinib in Participants With Moderate Hepatic Impairment Compared to Healthy Participants
Description: Maximum Plasma Concentration (Tmax) is defined as time of maximum observed plasma concentration and was calculated using non-compartmental analysis.
Time Frame: as for outcome 1
Population: Pharmacokinetic parameter was assessed using the Pharmacokinetic Analysis Set.
Measure: Mean (Full Range); unit: hours
Arm/Group | Normal HF | Moderate HI
Number analyzed (Participants) | 8 | 8
hours | 3.0 [2.5 to 4.5] | 10.0 [4.5 to 48.0]

11. Secondary Outcome: Area Under the Concentration-Time Curve (AUCinf) of of ZAAD-1006a Metabolite Following a Single Dose of Pexidartinib in Participants With Moderate Hepatic Impairment Compared to Healthy Participants
Description: Area Under the Concentration-Time Curve (AUCinf) is defined as area under the plasma concentration-time curve from the time of dosing extrapolated to infinity and AUClast is defined as AUC from time 0 to the last measurable concentration, as calculated by the linear up-log down trapezoidal method. AUCinf and AUClast are reported and were calculated using non-compartmental analysis.
Time Frame: as for outcome 1
Population: Pharmacokinetic parameters were assessed using the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng•h/mL
Arm/Group | Normal HF | Moderate HI
Number analyzed (Participants) | 8 | 8
ng•h/mL
  AUCinf | 43700 (29300) | 78100 (38300)
  AUClast | 42700 (28800) | 72700 (36900)

12. Secondary Outcome: Terminal Elimination Half-Life (t1/2) of ZAAD-1006a Metabolite Following a Single Dose of Pexidartinib in Subjects Participants With Moderate Hepatic Impairment Compared to Healthy Participants
Description: as for outcome 6
Time Frame: as for outcome 1
Population: Pharmacokinetic parameter was assessed using the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Normal HF | Moderate HI
Number analyzed (Participants) | 8 | 8
hours | 28.9 (4.03) | 37.9 (14.5)

13. Secondary Outcome: Metabolite-to-Parent Ratio (MPR) Corrected for Molecular Weight of ZAAD-1006a Metabolite Following a Single Dose of Pexidartinib in Participants With Moderate Hepatic Impairment Compared to Healthy Participants
Description: AUCinf is defined as area under the plasma concentration-time curve from the time of dosing extrapolated to infinity and AUClast is defined as AUC from time 0 to the last measurable concentration, as calculated by the linear up-log down trapezoidal method. MPR is defined as a metabolite to parent ratio with metabolite as the numerator and the parent as the denominator. MPR corrected for molecular weight of ZAAD-1006a of AUCinf and AUClast are reported and were calculated using non-compartmental analysis.
Time Frame: as for outcome 1
Population: Pharmacokinetic parameter was assessed using the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Normal HF | Moderate HI
Number analyzed (Participants) | 8 | 8
ratio
  MPR AUCinf | 1.08 (0.273) | 1.27 (0.405)
  MPR AUClast | 1.09 (0.275) | 1.30 (0.373)

14. Secondary Outcome: Percentage of Plasma Protein Binding of Pexidartinib and ZAAD-1006a Following a Single Dose in Participants With Moderate Hepatic Impairment Compared to Healthy Participants
Description: Protein binding (percentage bound) was determined in all participants at 2.5h and 24h post-dose. Plasma was harvested and analyzed for the quantification of pexidartinib using a validated liquid chromatography-tandem mass spectrometry method and the ZAAD-1006a metabolite was analyzed using a qualified liquid chromatography-tandem mass spectrometry assay.
Time Frame: 2.5 and 24 hours post-dose
Population: The pharmacokinetic parameter of Percentage of Plasma Protein Binding was assessed using the Pharmacokinetic Analysis Set. Only those participants with data available at the specified timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of protein binding
Arm/Group | Normal HF | Moderate HI
Number analyzed (Participants) | 8 | 8
percentage of protein binding
  Pexidartinib at 2.5hrs post-dose: number analyzed (Participants) | 7 | 8
  Pexidartinib at 2.5hrs post-dose | 99.9727 (0.00365) | 99.9695 (0.00454)
  Pexidartinib at 24hrs post-dose: number analyzed (Participants) | 6 | 8
  Pexidartinib at 24hrs post-dose | 99.9703 (0.00765) | 99.9664 (0.00815)
  ZAAD-1006a at 2.5hrs post-dose | 99.8605 (0.01056) | 99.8570 (0.03238)
  ZAAD-1006a at 24hrs post-dose | 99.8631 (0.02055) | 99.8534 (0.03868)

15. Secondary Outcome: Number of Participants Reporting Treatment-Emergent Adverse Events (TEAE) by System Organ Class and Preferred Term Following a Single Dose of Pexidartinib in Participants With Moderate Hepatic Impairment Compared to Healthy Participants
Description: A Treatment-Emergent Adverse Event (TEAE) is defined as any event not present prior to the initiation of the drug treatment or any event already present that worsens in either intensity or frequency following exposure to the drug treatment.
Time Frame: Post-dose and up to 30 days
Population: TEAEs were assessed using the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Normal HF | Moderate HI
Number analyzed (Participants) | 8 | 8
Participants
  Any TEAEs | 1 | 2
  Eye Disorders (Conjunctival haemorrhage) | 0 | 1
  Gastrointestinal Disorders (Dyspepsia) | 0 | 1
  Nervous System Disorders (Headache) | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the date of signing the informed consent form up to 30 days after last dose, up to 10 months.
Description: Adverse events were defined as any untoward, unfavorable, unintended medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. All-cause mortality includes all deaths that occurred during the study and within the 30 days after the last dose of the study drug.
Arm/Group | Normal HF | Moderate HI
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 1/8 | 2/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Normal HF (N=8) | Moderate HI (N=8)
Conjunctival haemorrhage (Eye disorders) | 0 | 1
Gastrointestinal disorders (Gastrointestinal disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-10): https://cdn.clinicaltrials.gov/large-docs/35/NCT04223635/Prot_SAP_000.pdf